CLINICAL TRIAL: NCT05812404
Title: A Randomized, Open-label, Three-period, Three-sequence, Multiple Dosing Crossover, Phase 1 Clinical Trial to Evaluate the Effect of DWP14012 on the Pharmacokinetics of DWC202201 After Co-administration of DWP14012 and DWC202201 in Healthy Subjects
Brief Title: Phase 1 Clinical Trial to Evaluate the Effect of DWP14012 on the Pharmacokinetics of DWC202201 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP14012109
Record Dates: First submitted 2022-11-14; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): * Treatment A: DWC202201 40 mg qd for 7 days
  * Treatment B: DWP14012 40 mg qd for 7 days, followed by DWC202201 40 mg qd + DWP14012 40 mg qd for 7 days
  * Treatment C: DWP14012 40 mg qd for 14 days
  Interventions: Drug: DWP14012; Drug: DWC202201
- Cohort 2 (Experimental): * Treatment C: DWP14012 40 mg qd for 14 days
  * Treatment A: DWC202201 40 mg qd for 7 days
  * Treatment B: DWP14012 40 mg qd for 7 days, followed by DWC202201 40 mg qd + DWP14012 40 mg qd for 7 days
  Interventions: Drug: DWP14012; Drug: DWC202201
- Cohort 3 (Experimental): * Treatment B: DWP14012 40 mg qd for 7 days, followed by DWC202201 40 mg qd + DWP14012 40 mg qd for 7 days
  * Treatment C: DWP14012 40 mg qd for 14 days
  * Treatment A: DWC202201 40 mg qd for 7 days
  Interventions: Drug: DWP14012; Drug: DWC202201

INTERVENTIONS:
Drug: DWP14012 — Potassium-competitive acid blocker
Drug: DWC202201 — Atorvastatin Calcium Trihydrate

SUMMARY:
A randomized, open-label, three-period, three-sequence, multiple dosing crossover, phase 1 clinical trial to evaluate the effect of DWP14012 on the pharmacokinetics of DWC202201 after co-administration of DWP14012 and DWC202201 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 50 years at screening
* Subjects with a body weight ≥ 50.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 kg/m2 to ≤ 27.0 kg/m2 at screening

  ※ BMI (kg/m2) = body weight (kg)/[height (m)]2
* Subjects who voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a sufficient explanation on this study and fully understanding the information
* Subjects who are eligible to participate in the study at the discretion of the investigator by physical examination, laboratory tests, and investigator questioning, etc.

Exclusion Criteria:

* Subjects with a disease or a history related to hepatobiliary system, kidney(severe kidney disorder ect.), nervous system, respiratory system, digestive system, endocrine system, hematology system, circulatory system(Heart failure, Torsades de pointes ect.), unrinary system, psychiatry ect.
* Subjects with digestive disease(gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal disease, Crohn's disease) or history of surgery(except appendectomy, hernia surgery) which can affect on saftey and pharmacodynamics
* Subjects with hypersensitivity or history of clinically significant hypersensitivity to drugs including potassium competitive acid blocker [P-CAB] class, aspirin, antibiotics, etc.
* Subjects with hereditary disorders including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.
* Subjects with history of inherited muscle disorders
* Subjects with a history of drug abuse or a positive result of using abusive drugs in the urine drug screen
* Subjects who participated in other clinical trials (including bioequivalence studies) within 6 months prior to the first scheduled dose of the IP
* Subjects who donated whole blood within 2 months, donated blood components within 1 month, or received blood transfusion within 1 month prior to the first scheduled dose
* Subjects who are unable to refrain from grapefruit-containing products from 3 days prior to the first scheduled dose until last discharge from hospital
* Subjects or their spouses or partners who are unable to use medically acceptable appropriate double-method of contraception or medically acceptable contraception throughout the study period and for at least 4 weeks after the last IP administration
* Subjects who are unable to refrain from smoking(>10pieces/day) from 3 days prior to the first scheduled dose until last discharge from hospital
* Subjects with alchoholic disorders or subjects who are unable to refrain from drinking(>21units/week) from 3 days prior to the first scheduled dose until last discharge from hospital
* Subjects who are unable to refrain from caffein(>5units/day) from 3 days prior to the first scheduled dose until last discharge from hospital

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-06-16 (Estimated)

PRIMARY OUTCOMES:
Atorvastatin Peak Plasma Concentration at steady state (Cmax,ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin Area under the plasma concentration versus time curve at steady state (AUCinf, ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]

SECONDARY OUTCOMES:
Atorvastatin Area under the plasma concentration extrapolated to infinity at steady state (AUC,ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin Time to peak drug concentration at staedy state (Tmax, ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin Terminal Half-life at steady state (T1/2,ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin Apparent total body clearance at steady state (CLss/F) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin Apparent volume of distribution at steady state (Vd,ss/F) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin active metabolite Area under the plasma concentration versus time curve at steady state (AUCinf, ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin active metabolite Terminal Half-life at steady state (T1/2,ss) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin active metabolite An estimate of the total body clearance at steady state (CL ss/F) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin active metabolite Apparent volume of distribution at steady state (Vd,ss/F) after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Atorvastatin active metabolite metabolic ratio after DWC202201 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Peak Plasma Concentration (Cmax) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan Area under the plasma drug concentration-time curve from 0 to tau (AUCtau) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan Area under the plasma drug concentration-time curve from 0 to infinity(AUCinf) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan The time of peak concentration (Tmax) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan Terminal Half-life (t1/2) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan Apparent Clearance (CL/F) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan Apparent Volume of Distribution After extravascular administration (Vd/F) after DWP14012 single dosing | [Time Frame: up to 64 days]
Fexuprazan Peak Plasma Concentration at steady state (Cmax,ss) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Area under the plasma drug concentration-time curve from 0 to tau at steady state (AUCtau,ss) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Area under the plasma drug concentration-time curve from 0 to infinity at steady state (AUCinf,ss) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Time of Maximum Concentration at steady state (Tmax,ss) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Terminal Half-life at steady state (t1/2,ss) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan An estimate of the total body clearance at steady state (CL ss/F) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Aapparent volume of distribution after extravascular administration at steady state (Vd,ss/F) after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan Accumulation ratio after DWP14012 multiple dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite Peak Plasma Concentration (Cmax) after single dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite Area under the plasma drug concentration-time curve from 0 to tau (AUCtau) after single dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite Area under the plasma concentration extrapolated to infinity (AUCinf) after single dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite The time of peak concentration (Tmax) after single dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite metabolic ratio after single dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite Peak Plasma Concentration at steady state (Cmax,ss) after multiple dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite AUCtau,ss AUCinf,ss Tmax,ss metabolic ratio | [Time Frame: up to 64 days]
Fexuprazan active metabolite Area under the plasma drug concentration-time curve from 0 to tau at steady state (AUCtau,ss) after multiple dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite Area under the plasma concentration extrapolated to infinity at steady state (AUCinf,ss) after multiple dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite The time of peak concentration at steady state (Tmax,ss) after multiple dosing | [Time Frame: up to 64 days]
Fexuprazan active metabolite metabolic ratio after multiple dosing | [Time Frame: up to 64 days]

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided